CLINICAL TRIAL: NCT05944991
Title: Effect of Olive Oil Massage on Growth in Preterm Low Birth Weight Neonate: A Randomized
Brief Title: Effect of Olive Oil Massage on Growth in Preterm Low Birth Weight Neonate: A Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Rumpa Mani Chowdhury, Dr.Rumpa Mani Chowdhury, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 11921
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Weight Gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olive oil message (Experimental): Give olive oil message 2 times per day
  Interventions: Other: Olive oil message

INTERVENTIONS:
Other: Olive oil message — Message of olive oil 2 times daily

SUMMARY:
STUDY TITLE: Effect of olive oil massage on growth of preterm low birth weight neonate: A randomized controlled clinical trial."

SUMMARY:

Preterm low birth weight (LBW) babies have more the risk of the neurological complications, physiological problems and mental retardation. Topical massage with natural oil is routinely practiced in some country. The positive effects of massage are weight gain, improved sleep/wake pattern, decreased the stress, early discharge from the neonatal intensive care unit (NICU), improve the skin integrity and enhanced parent's infant bonding. This randomized control trial study will be conducted in the Department of Neonatology,Bangabandhu Sheikh Mujib Medical University(BSMMU) and post natal ward of Department of Obstetrics and Gynecology with the aim to assess the effect of olive oil message on growth in low birth weight neonate. In this study tolal 50 inborn low birth weight neonate will be enrolled. Out of which 25 will be in intervention group and 25 will be in control group. In the intervention group, mothers will be encouraged to massage their babies with 10 ml of olive oil for 15 min, twice a day until 10 days of life. Those allocated to the control group were received care as usual. Weight and head circumference was measured at enrolment, after 10 days and on 30 days of age in both the groups. Comparisons between groups for categorical variables will be performed using the χ2-test. Student's t-test will be used to compare two groups for normally distributed quantitative data. The difference will be considered significant for P < 0.05.

DETAILED DESCRIPTION:
General Objective:

To observe the effect of Olive oil message on growth of preterm low birth weight babies.

Specific Objectives:

1. To measure the growth of preterm low birth weight neonate with or without olive oil message groups.
2. To measure the weight gain velocity of preterm low birth weight neonate with or without olive oil message groups.
3. To compare the growth and weight gain velocity between of two groups.

Study design: Randomized control trial.

Place of study: Department of Neonatology and Department of Obstetrics & Gynecology, Bangabandhu Sheikh Mujib Medical University (BSMMU), Shahbag, Dhaka, Bangladesh.

Study period: 6 months after IRB clearance. Study population: All preterm low birth weight neonate who will stay with mother in post-natal ward.

Inclusion Criteria:

1. Babies with 1500 to 2499 grams birth weight.
2. Age 24 to 48 hours.
3. Babies on full breast feed
4. Hemodynamically stable babies.

Exclusion criteria:

1. Newborns with multiple congenital anomalies
2. Preterm low birth weight neonate who required admission in NICU.
3. If there were symptoms such as fever, respiratory distress, muscle stiffness, vomiting.
4. Sensitivity to olive oil.

Main outcome variable: Growth of the neonate

Study procedure:

All eligible neonate will be selected as per inclusion and exclusion criteria. After explaining the aims of the study and signing an informed consent by the parents, the neonates will be divided into two groups by using a table of random numbers generated by the computer. Group A will be served as the control group, here babies in this group will be get kangaroo mother care, nothing applied to skin as per institutional protocol. Group B will receive message with olive oil along with other care as per institutional protocol. Details of obstetric history, mode of delivery, the socioeconomic status, and presence of risk factors for sepsis will be noted in predesigned proforma in both group.

Mathai et al, has described a standardised massage protocol which has been followed by most studies on massage therapy and adopted in this study also [21]. The Mathai's massage therapy consists of both tactile and kinesthetic stimulation.

Inborn low birth weight neonates from the ages of 2 days will be chosen for the study. Two massage sessions will be given in a day, each session for 15 minutes. Oil massage will be given for 30 days. Mothers will be taught the techniques through demonstration by trained residents and will be encouraged to massage their babies. The massage session will be initiated an hour after a feed to avoid regurgitation or vomiting of the feed. The infant in the intervention group will be given olive oil (same brand) massage with 5mL/kg of body weight being applied per session. During massage, the neonates will be placed completely naked on a plastic cover. The mother will be instructed to warm and lubricate her hands before starting of massage and to remain silent during intervention. If the baby started crying or passed urine or stools during the session it will temporarily stopped till the baby will comfortable again. The massage protocol is as follows.

Phase I: This will be done in the prone position. Twelve firm strokes with palms of the hands of 5 seconds each, were provided in each area as follows: (a) Head from forehead hairline over scalp down to neck with alternate hands; (b) Neck from midline outwards with both hands simultaneously; (c) Shoulders from midline outwards with both hands simultaneousously; and (d) Back from nape of neck down to buttocks with firm, long stroke with alternate hands.

Phase-II: This will be done in the supine position. Twelve firm stroke with palms of the hands, of 5 seconds each, were provided in each area as follows: (a) Forehead - From midline, outwards with both hands simultaneously; (b) Cheeks - From side of nose, with both hands simultaneously in rotating and clockwise direction for left cheek and anticlockwise direction for right cheek; (c) Chest- 'butterfly' stroking from midline upwards, outwards, downwards and inwards back to initiating point; (d) Abdomen - From the appendix, in a clock wise direction around abdomen avoiding the epigastrium and probes, with gentle strokes; (e) Upper limbs (each separately)- from shoulders to wrist using alternate hands for stroking; ( f ) Lower limbs (each separately) - from hips to ankles using alternate hands for stroking; (g) Palms - from wrist to finger tips using alternate hands for stroking; and (h) Soles- from heel to toe tips using alternate hands for stroking.

Phase-III: This will be done in the supine position and consisted of passive flexion and extension movements of the limbs at each large joint (shoulder, elbow, hip, knee and ankle) as 5 events of 2 seconds each in each area. Those will be allocated to the control group will be received care as usual.

The weight,length,OFC of LBW neonate in both the groups will be measured and recorded on day of start message,10 days after and at 30 days. Regular communication with mother will be continue when they will be at home over phone.

In this way the study will be conducted for a period of 6 months and the data will be collected, tabulated and analysed.Adverse effects due to the massage will also looked for.

.

ELIGIBILITY:
Inclusion Criteria:1. Babies with 1500 to 2499 grams birth weight. 2. Age 24 to 48 hours. 3. Babies on full breast feed 4.Hemodynamically stable babies.

-

Exclusion Criteria:

-1. Newborns with multiple congenital anomalies 2. Preterm low birth weight neonate who required admission in NICU. 3. If there were symptoms such as fever, respiratory distress, muscle stiffness, vomiting.

4. Sensitivity to olive oil.

Ages: 24 Hours to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Effect of olive oil massage on growth of preterm low birth weight neonate: A randomized controlled clinical trial." | 6 months
  To assess weight gain of preterm baby after olive oil message.

CONTACTS AND LOCATIONS:
Locations (1):
- BSMMU, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No